CLINICAL TRIAL: NCT02296853
Title: A Phase 1, Open-Label, Parallel-Group, Single Dose Study to Evaluate the Pharmacokinetics of Tenofovir Alafenamide (TAF) in Subjects With Normal Hepatic Function and Subjects With Severe Hepatic Impairment
Brief Title: Study to Evaluate the Pharmacokinetics of Tenofovir Alafenamide (TAF) in Adults With Normal Hepatic Function and Adults With Severe Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-320-1615; 2014-004426-18 (EudraCT Number)
Record Dates: First submitted 2014-11-18; First posted 2014-11-20 (Estimated); Results first posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-11

CONDITIONS: Hepatitis B Virus
Keywords: Severe Hepatic Impairment
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Severe Hepatic Impairment Group (Experimental): Participants with severe hepatic impairment will receive a single oral dose of TAF 25 mg on Day 1.
  Interventions: Drug: TAF
- Matched Normal Hepatic Function Group (Active Comparator): Participants with normal hepatic function will receive a single oral dose of TAF 25 mg on Day 1.
  Interventions: Drug: TAF

INTERVENTIONS:
Drug: TAF — 25 mg tablet administered orally

SUMMARY:
The primary objective of this study is to evaluate the single-dose pharmacokinetics of tenofovir alafenamide (TAF) and its metabolite tenofovir (TFV) in participants with normal hepatic function and in participants with severe hepatic impairment.

ELIGIBILITY:
Key Inclusion Criteria:

* Screening laboratory parameters within defined thresholds
* Creatinine clearance must be ≥ 60 mL/min

Key Exclusion Criteria:

* Females who are pregnant or nursing or males who have a pregnant partner
* Infection with hepatitis B virus (HBV) or HIV
* History of clinically significant illness (including psychiatric or cardiac) or any other medical disorder that may interfere with participant treatment and/or adherence to the protocol

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-12-22 (Actual); Primary Completion 2015-04-17 (Actual); Study Completion 2015-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (5):
- United States (3):
  - Miami, Florida
  - Orlando, Florida
  - San Antonio, Texas
- Munich, Germany
- Gratton, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Germany, New Zealand, and the United States. The first participant was screened on 22 December 2014. The last study visit occurred on 17 April 2015.
Pre-assignment Details: 28 participants were screened.
Groups:
- Severe Hepatic Impairment Group: Participants with severe hepatic impairment received a single oral dose of tenofovir alafenamide (TAF) 25 mg on Day 1.
- Matched Normal Hepatic Function Group: Participants with normal hepatic function received a single oral dose of TAF 25 mg on Day 1.
Period: Overall Study
Arm/Group | Severe Hepatic Impairment Group | Matched Normal Hepatic Function Group
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all enrolled participants who received at least 1 dose of study drug.
Groups:
- Severe Hepatic Impairment Group: Participants with severe hepatic impairment received a single oral dose of TAF 25 mg on Day 1.
- Total: Total of all reporting groups
Arm/Group | Severe Hepatic Impairment Group | Matched Normal Hepatic Function Group | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (7.3) | 55 (9.3) | 56 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 7 | 6 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 10 | 9 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 1 | 3 | 4
  New Zealand | 2 | 2 | 4
  United States | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic (PK) Parameter: AUCinf of Tenofovir Alafenamide (TAF), Its Metabolite Tenofovir (TFV) and Free (Unbound) TAF
Description: AUCinf is defined as the concentration of drug extrapolated to infinite time.
Time Frame: Predose (≤5 minutes), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 8, 12, 24, 36, 48, 60, 72, 96, 120, and 144 hours postdose on Day 1
Population: Participants in the PK Analysis Set (consisted of all enrolled participants who received at least 1 dose of the study drug and had at least 1 non-missing PK concentration data for each respective analyte) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Severe Hepatic Impairment Group | Matched Normal Hepatic Function Group
Number analyzed (Participants) | 10 | 8
h*ng/mL
  TAF | 120.6 (33.96) | 228.2 (85.30)
  TFV | 219.9 (118.70) | 304.0 (72.45)
  Free (unbound) TAF | 42.8 (11.76) | 46.5 (17.78)
Statistical Analysis 1: Comparison: Severe Hepatic Impairment Group vs Matched Normal Hepatic Function Group; TAF: Severe Hepatic Impairment Group vs. Matched Normal Hepatic Function Group; Test type: Equivalence — Sample size calculations were done in Query Advisor 6.0 by using the "Two-group t-test of equal means (equal n's)" module with α (one-sided) = 0.05, upper equivalence limit = ln(2.0) = 0.691, and expected difference = 0; GLSM ratio percentage = 54.04, 90% CI 2-sided [41.98 to 69.56] — Here, GLSM is geometric least square mean
Statistical Analysis 2: Comparison: Severe Hepatic Impairment Group vs Matched Normal Hepatic Function Group; TFV: Severe Hepatic Impairment Group vs. Matched Normal Hepatic Function Group; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; GLSM ratio percentage = 63.06, 90% CI 2-sided [42.90 to 92.70]
Statistical Analysis 3: Comparison: Severe Hepatic Impairment Group vs Matched Normal Hepatic Function Group; Free (unbound) TAF: Severe Hepatic Impairment Group vs. Matched Normal Hepatic Function Group; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; GLSM ratio percentage = 94.42, 90% CI 2-sided [72.48 to 122.99]

2. Primary Outcome: PK Parameter: Cmax of TAF, Its Metabolite TFV and Free (Unbound) TAF
Description: Cmax is defined as the maximum concentration of drug.
Time Frame: as for outcome 1
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Severe Hepatic Impairment Group | Matched Normal Hepatic Function Group
Number analyzed (Participants) | 10 | 10
ng/mL
  TAF | 79.6 (39.31) | 176.0 (79.77)
  TFV | 7.5 (3.95) | 7.6 (1.83)
  Free (unbound) TAF | 29.9 (17.36) | 36.2 (18.38)
Statistical Analysis 1: Comparison: Severe Hepatic Impairment Group vs Matched Normal Hepatic Function Group; TAF: Severe Hepatic Impairment Group vs. Matched Normal Hepatic Function Group; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; GLSM ratio percentage = 45.10, 90% CI 2-sided [31.66 to 64.25]
Statistical Analysis 2: Comparison: Severe Hepatic Impairment Group vs Matched Normal Hepatic Function Group; TFV: Severe Hepatic Impairment Group vs. Matched Normal Hepatic Function Group; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; GLSM ratio percentage = 89.88, 90% CI 2-sided [64.77 to 124.72]
Statistical Analysis 3: Comparison: Severe Hepatic Impairment Group vs Matched Normal Hepatic Function Group; Free (unbound) TAF: Severe Hepatic Impairment Group vs. Matched Normal Hepatic Function Group; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Sample size calculations were done in Query Advisor 6.0 by using the "Two-group t-test of equal means (equal n's)" module with α (one-sided) = 0.05, upper equivalence limit = ln(2.0) = 0.691, and expected difference = 0; GLSM ratio percentage = 82.16, 90% CI 2-sided [56.58 to 119.31]

3. Primary Outcome: PK Parameter: AUClast of TAF, Its Metabolite TFV and Free (Unbound) TAF
Description: AUClast is defined as the concentration of drug from time zero to the last observable concentration.
Time Frame: as for outcome 1
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Severe Hepatic Impairment Group | Matched Normal Hepatic Function Group
Number analyzed (Participants) | 10 | 10
h*ng/mL
  TAF | 113.1 (30.85) | 225.7 (85.09)
  TFV | 184.2 (99.86) | 256.7 (59.91)
  Free (unbound) TAF | 41.7 (11.17) | 46 (17.75)
Statistical Analysis 1: Comparison: Severe Hepatic Impairment Group vs Matched Normal Hepatic Function Group; TAF: Severe Hepatic Impairment Group vs. Matched Normal Hepatic Function Group; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; GLSM ratio percentage = 51.20, 90% CI 2-sided [40.11 to 65.36]
Statistical Analysis 2: Comparison: Severe Hepatic Impairment Group vs Matched Normal Hepatic Function Group; TFV: Severe Hepatic Impairment Group vs. Matched Normal Hepatic Function Group; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; GLSM ratio percentage = 62.04, 90% CI 2-sided [41.92 to 91.82]
Statistical Analysis 3: Comparison: Severe Hepatic Impairment Group vs Matched Normal Hepatic Function Group; Free (unbound) TAF: Severe Hepatic Impairment Group vs. Matched Normal Hepatic Function Group; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; GLSM ratio percentage = 93.28, 90% CI 2-sided [72.62 to 119.8]

4. Secondary Outcome: Percentage of Participants Experiencing Treatment-Emergent Adverse Events (TEAEs)
Description: TEAEs are events that meet one of the following criteria: any AEs with onset date of on or after the study drug start date and no later than 30 days after permanent discontinuation of study drug or any AEs leading to premature discontinuation of study drug.
Time Frame: Day 1 plus 30 days
Population: The Safety Analysis Set included all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Severe Hepatic Impairment Group | Matched Normal Hepatic Function Group
Number analyzed (Participants) | 10 | 10
percentage of participants | 40.0 | 30.0

5. Secondary Outcome: Percentage of Participants Experiencing Treatment Emergent Laboratory Abnormalities
Description: Treatment-emergent laboratory abnormalities were defined as values that increase at least one toxicity grade from baseline. These were graded as Grade 1: mild, Grade 2: moderate, Grade 3: severe, Grade 4: life-threatening. The most severe graded abnormality from all tests was counted for each participant.
Time Frame: Day 1 plus 30 days
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Severe Hepatic Impairment Group | Matched Normal Hepatic Function Group
Number analyzed (Participants) | 10 | 10
percentage of participants
  Grade 1 | 40.0 | 30.0
  Grade 2 | 40.0 | 30.0
  Grade 3 | 20.0 | 10.0
  Grade 4 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 plus 30 days
Description: The Safety Analysis Set included all enrolled participants who received at least 1 dose of study drug.
Groups:
- Matched Normal Hepatic Function Group: Participants with normal hepatic function received a single oral dose of TAF 25 mg of on Day 1.
Arm/Group | Severe Hepatic Impairment Group | Matched Normal Hepatic Function Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/10
Other Adverse Events (participants affected / at risk) | 4/10 | 3/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Severe Hepatic Impairment Group (N=10) | Matched Normal Hepatic Function Group (N=10)
Hepatic failure (Hepatobiliary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Severe Hepatic Impairment Group (N=10) | Matched Normal Hepatic Function Group (N=10)
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years